CLINICAL TRIAL: NCT00824811
Title: A Double-Blind Study Evaluating the Safety and Efficacy of Cyclosporine Ophthalmic Emulsion 0.05% [Restasis] in Subjects With Epiphora Secondary to Docetaxel [Taxotere] Treatment for Various Cancers
Brief Title: Topical Cyclosporine vs. Placebo for Epiphora Associated With Docetaxel
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual.
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2007-0757
Record Dates: First submitted 2009-01-16; First posted 2009-01-19 (Estimated); Last update posted 2012-08-02 (Estimated); Status verified 2012-08

CONDITIONS: Epiphora
Keywords: Epiphora; Breast Cancer; Lung Cancer; Prostate Cancer; Non-small cell lung cancer; Bladder Cancer; Esophageal Cancer; Head and Neck Cancer; HNC; Small Cell Lung Cancer; SCLC; Ovarian Cancer; Stomach Cancer; Canalicular Stenosis; Excessive tearing; Eye inflammation; Cyclosporine Ophthalmic Emulsion 0.05%; Docetaxel; Taxotere; Restasis®; Cyclosporine; Cyclosporine eye drops; FML Forte®; Fluorometholone 0.25% ophthalmic suspension; Fluorometholone eye drops; Fluorometholone; Refresh Endura™; Lubricant eye drops; Eye drops
MeSH Terms: conditions — Lacrimal Apparatus Diseases; Breast Neoplasms; Lung Neoplasms; Prostatic Neoplasms; Carcinoma, Non-Small-Cell Lung; Urinary Bladder Neoplasms; Esophageal Neoplasms; Head and Neck Neoplasms; Small Cell Lung Carcinoma; Ovarian Neoplasms; Stomach Neoplasms; Lacerations; Endophthalmitis | interventions — Cyclosporins; Lubricant Eye Drops; Fluorometholone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1: Cyclosporine eye drops (Experimental): Cyclosporine Eye Drops (Restasis) 1 drop twice/day for 84 days to both eyes + Fluorometholone Eye Drops (FML Forte) on declining dose schedule.
  Interventions: Drug: Cyclosporine Eye Drops (Restasis); Drug: Fluorometholone Eye Drops (FML Forte®)
- Group 2: Lubricant Eye Drops (Experimental): Lubricant Eye Drops (Refresh Endura) 1 drop twice/day for 84 days to both eyes + Fluorometholone Eye Drops (FML Forte) on declining dose schedule.
  Interventions: Drug: Lubricant Eye Drops (Refresh Endura™); Drug: Fluorometholone Eye Drops (FML Forte®)

INTERVENTIONS:
Drug: Cyclosporine Eye Drops (Restasis) — One drop twice a day (approximately 12 hours between instillations) for 84 consecutive days to both eyes.
  Other Names: Cyclosporine eyedrops; Cyclosporine Opthalmic Emulsion 0.05%
  Arms: Group 1: Cyclosporine eye drops
Drug: Lubricant Eye Drops (Refresh Endura™) — One drop twice a day (approximately 12 hours between instillations) for 84 consecutive days to both eyes.
  Other Names: Refresh Endura™ eye drops
  Arms: Group 2: Lubricant Eye Drops
Drug: Fluorometholone Eye Drops (FML Forte®) — Week 1: One drop four times a day to both eyes.
  Week 2: One drop three times a day to both eyes.
  Week 3: One drop twice a day to both eyes.
  Week 4: One drop once a day to both eyes.
  Wait at least 10 minutes after Restasis® or Refresh Endura™ instillation to instill FML Forte®.
  Other Names: Fluorometholone 0.25% Opthalmic Suspension

SUMMARY:
Objective:

To evaluate the safety and efficacy of topical cyclosporine eye drops (Restasis®) for the treatment of epiphora caused by canalicular stenosis secondary to Docetaxel (Taxotere®) treatment for various cancers.

DETAILED DESCRIPTION:
The Study Drugs:

Restasis® is also known as cyclosporine ophthalmic emulsion 0.05% (cyclosporine eye drops). It is designed to decrease eye inflammation.

FML Forte® is also known as fluorometholone 0.25% ophthalmic suspension (fluorometholone eye drops). It is designed to decrease eye inflammation. Fluorometholone eye drops are commonly used to help to control epiphora.

In this study, an additional type of eye drops will be used for comparison with cyclosporine eye drops. This second type of eye drops is called Refresh Endura™ (lubricant eye drops), which is designed to relieve dry eyes. Unlike cyclosporine and fluorometholone, it does not have active ingredients designed to treat epiphora.

Study Groups:

If you are found to be eligible to take part in this study, you will be assigned to 1 of 2 groups. The way of assigning participants to groups is mostly random, as in the flip of a coin. However, your epiphora score (how often you dabbed your tears, as recorded in a diary) will also affect what group you are assigned to.

Group 1 will receive cyclosporine eye drops and fluorometholone eye drops. Group 2 will receive lubricant eye drops and fluorometholone eye drops.

Neither you nor the study staff will know whether you are receiving cyclosporine eye drops or lubricant eye drops. However, if needed for your safety, the study staff will be able to find out which one you are receiving.

Study Drug Administration Your first dose of the study drugs will be given in the clinic on Day 1. After that, you will give yourself the rest of the doses at home. The study staff will teach you how to use the eye drops, and you will be given written instructions. Study data will be collected on both eyes, and you will apply the drops to both eyes.

If you wear contact lenses, be sure to take your contact lenses out before using the eye drops. Fifteen (15) minutes after your dose of the eye drops, you may put your contact lenses back in.

If you are in Group 1, you will apply 1 drop of cyclosporine eye drops to each eye, 2 times a day, for 84 days (12 weeks) in a row. You should wait about 12 hours between doses.

If you are in Group 2, you will apply 1 drop of lubricant eye drops to each eye, 2 times a day, for 84 days in a row. You should wait about 12 hours between doses.

All study participants must wait at least 10 minutes after you have applied your other eye drops (cyclosporine or the lubricant) before you can apply the fluorometholone eye drops.

All study participants will receive fluorometholone eye drops. During Week 1, you will apply 1 drop to each eye, 4 times a day. During Week 2, you will apply 1 drop to each eye, 3 times a day. During Week 3, you will apply 1 drop to each eye, 2 times a day. During Week 4, you will apply 1 drop to each eye, once a day.

Study Visits:

On Visit 1 (Day -1 or -2), your eye doctor and/or study staff will ask you to sign the written informed consent. Screening tests will be done, which include urine pregnancy test for all women who are able to become pregnant, and other eye exams, such as Best Corrected Visual Acuity, Biomicroscopy, Intraocular Pressure (IOP), Epiphora Assessments, Schirmer's Test, and Probing and Irrigation Test. Your eye doctor and/or assistant will explain these different eye exams, or any questions you may have, at the day of your visit. You will also be asked about the different medications that you are currently taking. You will be given participant diaries for you to record or keep track of your medication use and how many times you dab your tears. You will then be given the schedule of your next visit.

On Visit 2 (Day 0 or baseline), the study staff will record how well you tolerate the study drugs and any side effects that may occur after the doses. You will also complete 2 questionnaires. The first questionnaire asks about the quality of your life and the second questionnaire asks about any problems with your vision that you may be experiencing. In total, they should take about 10-15 minutes to complete.

You will be given additional patient diaries. In the first diary, you will record any missed doses of the study drugs. In the second diary, you will record how many times you dab tears from your eyes and/or face, starting 24 hours before each clinic visit.

You should bring the completed patient diaries and the used containers of the study drugs with you to every study visit.

At Weeks 2, 4, and 8, the following procedures will be performed:

* You will have a routine eye exam to check the status of the epiphora. The same eye tests will be performed as at screening. However, the routine procedure called "probing and irrigation" (a test of the tear ducts, involving water) may not need to be repeated. The probing and irrigation procedure will only be performed if the epiphora seems to have gotten worse. In that case, the probing and irrigation procedure will help the doctor decide whether to recommend that you consider additional treatments.
* You will be asked about any side effects you may have experienced, any other drugs or treatments you may be receiving, and any other changes to your current drugs or treatments.
* You will repeat the quality-of-life questionnaire. You will also complete a second questionnaire about your overall eye comfort and a third questionnaire about the eye tearing symptoms. In total, these questionnaires should take about 20 minutes to complete.

Length of Study Participation:

You may stay on study treatment for up to 12 weeks. If intolerable side effects occur, or the epiphora gets worse and the study doctor thinks you should consider surgery to treat it, you will be taken off study treatment early.

End-of-Study Visit:

After your last dose of the study drugs (at Week 12, or earlier if you go off study treatment early), you will return for an end-of-study visit. At this visit, the following procedures will be performed:

* You will have the same procedures performed as at Weeks 2, 4, and 8.
* You will complete the quality-of-life questionnaire, the questionnaire that asks about any problems with your vision, and the questionnaire that asks if your eye tearing symptoms have improved or gotten worse compared to the days before you started the study. In total, these questionnaires should take about 20 minutes to complete.
* Women who are able to have children will have a urine pregnancy test.

THIS IS AN INVESTIGATIONAL STUDY. Cyclosporine eye drops, fluorometholone eye drops, and Refresh Endura™ lubricant eye drops are commercially available for other eye conditions. They are not FDA approved for use in treating epiphora. At this time and for this purpose, they are considered experimental. This includes fluorometholone eye drops, which are commonly used to treat epiphora but are not FDA approved for this use.

Up to 40 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. male or female subjects 18 years of age or older in good general health;
2. provide verbal and written informed consent as well as written release of health and study information;
3. clinically diagnosed by the investigator to have mild to severe epiphora [grades 2, 3 or 4 on a five-point scale (0-4)] in one or both eyes;
4. diagnosed with any of the following types of cancer: breast, non-small cell lung, prostate, bladder, esophageal, head and neck, small cell lung, ovarian and stomach;
5. experiencing symptoms of epiphora after receiving Docetaxel (Taxotere®) at the frequency of at least every 3 weeks for his/her cancer;
6. must have less than grade II canalicular stenosis on probing and irrigation at baseline;
7. following a prescribed course of Docetaxel (Taxotere®) and accommodating this course without excessive allergic reaction, nausea and/or other adverse reaction (mild or otherwise);
8. expected to remain on Docetaxel (Taxotere®) therapy for at least 4 weeks after enrollment in the study;
9. women of childbearing potential must be willing to practice effective contraception for the duration of the study (i.e. abstinence, spermicide, condoms, or birth control pills [BCP]); {NOTE: Females on birth control pills (BCP) must be stable on the same type and dose of pill for at least three months prior to entering the study and must not change the type of BCP or dosing regimen during the study. Those who have used BCPs in the past must have discontinued usage at least 3 months prior to the start of the study}
10. women of child bearing potential must have a negative urine pregnancy test at the screening visit and must not be lactating; and
11. willing and able to instill the study medications as directed, comply with study instructions and return to the clinic for required visits.

Exclusion Criteria:

1. experiencing excessive allergic reaction;
2. receiving any medications which may interfere with Docetaxel (Taxotere®) treatment for subject's cancer;
3. experiencing any concomitant disease which might interfere with the diagnosis and treatment of epiphora
4. changed their hormone replacement or deprivation therapy (i.e., estrogen replacement or estrogen and androgen deprivation) program within three months of the baseline/screening visit or anticipate starting such a program during the course of the study;
5. anticipated contact lens wear during any portion of the study;
6. changed their treatment regimen of beta blocking agents, or cholinergic agonists within three months of the baseline/screening visit or anticipate changing, starting, or ending such a regimen during the course of the study;
7. use of ocular ointments (including over-the-counter ointments) within one week of the baseline/screening visit;
8. used topical (including ophthalmic) or systemic cyclosporine within 90 days of the baseline/screening visit;
9. diagnosed with acne rosacea and currently on any systemic tetracycline antibiotic or any other prescribed treatment such as metronidazole, or have used any prescribed treatment for acne rosacea in the past;
10. active ocular infection or inflammation in any eye;
11. active ocular allergy in any eye;
12. abnormal dilated fundus examination indicative of intraocular tumor presence;
13. corneal disorder or abnormality that affects cornea sensitivity or normal spreading of the tear film in any eye;
14. severe blepharitis or obvious inflammation of the lid margin in any eye which, in the judgment of the investigator, may interfere with the interpretation of the study results;
15. history of punctal occlusion, canalicular stenosis or nasolacrimal duct blockage.
16. unable to cannulate the puncta (grade 3 on the Canalicular Stenosis Scale);
17. unable to successfully irrigate the canaliculi;
18. Schirmer's Test - Standard Test (with anesthesia) result of </= 3 mm;
19. epiphora is due to reflex tearing resulting from dry eye syndrome;
20. history of anterior segment surgery or trauma in either eye which would affect corneal sensitivity (e.g., cataract surgery, Photorefractive keratectomy (PRK), Laser-Assisted Sub-Epithelial Keratectomy (or Laser Epithelial Keratomileusis) (LASEK/LASIK) or any surgery involving a limbal or corneal incision) within the last 12 months;
21. current use, use within 2 weeks prior to Day 0 (baseline) or likely to use during the study period of any topical ophthalmic medications (e.g., antibiotics, glaucoma medications) other than ophthalmic medications used in this study;
22. known allergy or hypersensitivity to Restasis® (cyclosporine A) and its excipients and/or FML Forte® (Fluorometholone 0.25%) and its excipients;
23. requirement for concomitant procedure(s)/therapy that would interfere with study objectives must cease use at least 4 weeks prior to enrollment and remain free from use of these procedures/therapies throughout duration of this study;
24. pregnant, nursing, or planning a pregnancy during the course of the study and females of childbearing potential, not using a reliable means of contraception;
25. clinically diagnosed by the investigator to have none to trace epiphora [grades 0 or 1on a five-point scale (0-4)] in either eye;
26. history of allergy or sensitivity to the other medications used in this study (Refresh Endura™) or their excipients;
27. history of herpetic eye disease;
28. any condition or situation which, in the investigator's opinion, may put the subject at significant risk, may confound the study results, or may interfere significantly with the subject's participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-06

PRIMARY OUTCOMES:
Patient Epiphora Grade Scores | Evaluated at Day 0 (Baseline) through Week 12
  Epiphora score (how often dabbed tears, as recorded in a diary) assessed on a five-point scale to grade epiphora: 0: None; 1: Trace; 2: Mild; 3: Moderate; 4: Severe. It is evaluated at Day 0, Weeks 2, 4, 8 and 12. The within-arm comparison made between baseline (Day 0) and Week 4.

CONTACTS AND LOCATIONS:
Overall Officials: Bita Esmaeli, MD, Principal Investigator — M.D. Anderson Cancer Center

REFERENCES:
- See also: The University of Texas M.D.Anderson Cancer Center — http://www.mdanderson.org